CLINICAL TRIAL: NCT05507775
Title: Digoxin for the Reinduction of Radioiodine Uptake in Metastatic or Locally Advanced Non-medullary Thyroid Carcinoma
Acronym: DIGUP-TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-500477-14-00
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Non-Medullary Thyroid Carcinoma
Keywords: Thyroid cancer; Digoxin; Autophagy; Redifferentiation; Radio-iodine refractory
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms | interventions — Digoxin

STUDY DESIGN:
Intervention Model Description: 10 participants with radioiodine refractory metastatic or locally advanced non-medullary thyroid carcinoma will enroll in this study. All participants will be treated according to the same protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with digoxin (Experimental): This arm will consist of 10 patients with radioiodine refractory non-medullary thyroid carcinoma. All participants will be treated according to the same protocol.
  Interventions: Drug: Digoxin tablet

INTERVENTIONS:
Drug: Digoxin tablet — Participants will be treated with digoxin tablets for 3 weeks. On the first they, participants will start with a starting dosage of 3x0.25mg with 6 hours between each administration. Thereafter they will continue with a dosage of 1x0.25mg. Participants aged >70 years or with body weight <55kg will initiate a starting dosage of 3x0.125mg with 6 hours between each administration. Thereafter they will continue with a dosage of 1x0.125mg.
  After one week the blood concentration of digoxin will be measured. According to this blood concentration, the dose of digoxin will be adjusted.

SUMMARY:
Non-medullary thyroid carcinoma has a good prognosis in most patients. However, a small subset of patients nevertheless develop metastatic or locally advanced and unresectable disease which in some cases also becomes radioiodine refractory. In these patients treatment options are very limited. Earlier cell line and animal studies have shown that digoxin can reinduce radioiodine uptake in non-medullary thyroid cancer. This study serves as a proof of principle study to assess the possibility of digoxin to reinduce radioiodine uptake in adult humans with metastatic or locally advanced non-medullary radioiodine refractory thyroid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Non-medullary thyroid carcinoma
* Having undergone total thyroidectomy and at least 1 treatment with [131]sodium iodine (NaI)
* Presence of local or metastatic disease, radiologically proven. A minimum of 1 target lesion (at least 1cm for soft tissue and 1.5cm for lymph nodes) must be present.
* Radioiodine refractory disease; at least one lesion without therapeutic relevant uptake at previous post-therapeutic scintigraphy and/or negative diagnostic [123]NaI-scan.
* The target lesion must not be eligible for local treatments.
* Hematologic lab values should be at least: absolute neutrophil count >1.4x10^9/liter, hemoglobin>5.5mmol/liter, thrombocytes >99x10^9/liter

Exclusion Criteria:

* Creatinine clearance <50ml/min and/or active kidney disease
* Cardiac arrhythmias
* Electrolyte disorder
* Concomitant drugs that interfere with digoxin metabolism such as P-glycoprotein inductors or inducers, including but not limited to penicillamine, sulfasalazin, tipranavir, amiodarona, diltiazem, itraconazole, ketoconazole, kinidin, lapatinib, propafenon, vemurafenib, verapamil, azithromycin, clarithromycin, erythromycin, roxithromycin, chloroquin, ciclosporin, anti hepatitis C drugs, anti-HIV drugs, hydroxychloroquine.
* Pregnancy, lactating or breast-feeding women.
* Having undergone a procedure with iodine contrast agent within the last 3 months.
* Prior therapy with radioactive iodine <6 months prior to participation.
* External beam radiation therapy <4 weeks prior to participation.
* Having undergone chemotherapy or targeted therapy <4 weeks prior to participation.
* Eastern Cooperative Oncology Group (ECOG) score >2.
* Use of other investigational drugs within 4 weeks preceding the first dose of digoxin treatment.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to digoxin.
* Uncontrolled intercurrent illness that would limit compliance with the study requirements.
* Unwillingness or inability to comply with study and follow-up procedures.
* Other active malignancies other than basal cell carcinoma. Malignancies that have been in complete remission over 2 years are not considered active malignancies.
* Rapidly progressive disease in which urgent start with systemic therapy is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Reinduction of radioiodine uptake in target lesion | 3 weeks
  At baseline and after 3 weeks of digoxin treatment, a scintigraphy scan will be conducted. Reinduction of radioiodine uptake is defined as enough uptake that a treatment with high-dose radioactive iodine is possible.

SECONDARY OUTCOMES:
Beneficial effects of high-dose radioactive iodine treatment after reinduction | 6 months
  Participants with reinduction of radioiodine uptake in the target lesion will be offered a treatment with high-dose radioactive iodine, according to the guidelines for the treatment of thyroid carcinoma. The beneficial effects of this treatment will be measured after 6 months with a computertomography scan and will be described using the RECIST criteria.
Safety of digoxin treatment | 3 weeks
  All serious adverse events (SAE) occuring during the digoxin treatment will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No